CLINICAL TRIAL: NCT03640039
Title: Comparative Study Evaluating Stability of Fracture Segments After Treatment of Mandibular Angle Fracture With 3d Strut Plate in Two Groups One With IMMF and Anthor Without IMMF ;Randomized Clinical Trial.
Brief Title: Comparative Study Evaluating Stability of Fracture Segments After Treatment of Mandibular Angle Fracture With 3d Strut Plate With or Without IMMF.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Khater tarek, Assistant lecturer., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2972018
Record Dates: First submitted 2018-07-29; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Mandible Fracture
Keywords: 3d strut plate; mandibular angle fracture
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Intervention Model Description: * A Radomized clinical trial.
  * Parallel group study.
  * A trial will be carried out in hospital of oral and maxillofacial surgery department - faculty of dentistry cairo university.
  * Equal randomization: participants with equal probabilities for intervention.
  * Positive controlled: both groups receiving treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group: 3d strut plate fixation without post op IMMF. (Experimental): Open reduction and internal fixation with 3d strut plate without post operative IMMF.
  Interventions: Procedure: 3d strut plate.
- control group: 3d srut plate fixation with post op IMMF. (Active Comparator): Open reduction and internal fixation with 3d strut plate with post operative IMMF for 15 days.
  Interventions: Procedure: 3d strut plate.

INTERVENTIONS:
Procedure: 3d strut plate. — Under general anathesia fracture will be exposed and fixed with 3d srut plate.Wound closed in standered fashion. patient will be released from operating room with out IMMF.

SUMMARY:
comparative study evaluating stability of fracture segments in mandibular angle fracture with 3d strut plate with or with out post operative IMMF.

DETAILED DESCRIPTION:
Two group of patient with mandibular angle fracture indicated for open reduction and internal fixation ,first group will be fixed with 3d stut plate with post operative IMMF. Second group will be fixed with 3d strut plate with out post operative IMMF.

Eligble patients will be randomised in equal proportions between study group (3d strut plate with out post operative IMMF) and control group (3d strut plate with post operative IMMF).

A- 3D strut plate without post operative IMMF:

* Pre operative computed tomography will be done for patient.
* Intra operative :all cases will under go general anathesia.
* Exposure of the fracture segments using vestubular incision.
* Inter-maxillary fixation will be done.
* The fracture segment will be reduced in normal anatomic postion guided with occlusion.
* The fracture segment will be fixed in postion using 3d srut plate.
* Closure of surgical incision.
* Post operative computed tomograghy will be done for the patient.
* Patient will be dismissed from operation room without IMMF.

B- 3D strut with post operative IMMF:

* Pre operative computed tomography will be done for patient.
* Intra operative :all cases will under go general anathesia.
* Exposure of the fracture segments using vestubular incision.
* Inter-maxillary fixation will be done.
* The fracture segment will be reduced in normal anatomic postion guided with occlusion.
* The fracture segment will be fixed in postion using 3d srut plate.
* Closure of surgical incision.
* Post operative computed tomograghy will be done for the patient.
* Patient will be dismissed from operation room with IMMF for 15 days.

Follow up for both groups :

Clinical examination will be done at first week post operative and patients will be examined every week for one month. Last follow up visit will be after three months post operative.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mandibular angle fracture with or witout other fracture indicated for Open reduction internal fixation in the mandible.
* Patient over 15 years old age and both sexes were included in this study.
* Patients should be free from any systemic disease that may affect normal healing of bone, and predictable outcome.
* Patients with good general condition allowing major surgical procedure under general anesthesia.
* Patients with physical and psychological tolerance.

Exclusion Criteria:

* Patients with comminuted fractures as it is not indicated for compression osteosynthesis like3d strut plate .
* Patients with high risk systemic diseases like uncontrolled diabetes mellitus. As uncontrolled diabetes mellitus has a negative impact on normal bone healing.
* Patients with old and/or mal-union fractures. As they will affect accuracy of reduction of the fractured segments.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-01-11 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
stability of fracture segments. | 15 days post operative.
  post operative bimanual manipulation of the fracture segment.

SECONDARY OUTCOMES:
inferior alveolar nerve injury. | pre operative and 1 week post operative.
  measurment by:Neurosensory testing: patient will be asked if there was numbness without stimulus and on stroking the lower lip skin with afinger.The patient will be asked to grade the sensation present on an analog scale from 0 (no sensation) to 10 (completely normal sensation)
Accuracy of fracture reduction. | one week post operative.
  Post operative. Through computed tomography by measuring inter ramus distance using lingula as reference to measure.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham A Hakam, Prof, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kellman RM. Repair of mandibular fractures via compression plating and more traditional techniques: a comparison of results. Laryngoscope. 1984 Dec;94(12 Pt 1):1560-7. PMID 6503575
- [Background] Saman M, Kadakia S, Ducic Y. Postoperative maxillomandibular fixation after open reduction of mandible fractures. JAMA Facial Plast Surg. 2014 Nov-Dec;16(6):410-3. doi: 10.1001/jamafacial.2014.543. PMID 25232835
- [Background] Guimond C, Johnson JV, Marchena JM. Fixation of mandibular angle fractures with a 2.0-mm 3-dimensional curved angle strut plate. J Oral Maxillofac Surg. 2005 Feb;63(2):209-14. doi: 10.1016/j.joms.2004.03.018. PMID 15690289
- [Background] Farmand M. [Experiences with the 3-D miniplate osteosynthesis in mandibular fractures]. Fortschr Kiefer Gesichtschir. 1996;41:85-7. German. PMID 8755408
- [Background] Vineeth K, Lalitha RM, Prasad K, Ranganath K, Shwetha V, Singh J. "A comparative evaluation between single noncompression titanium miniplate and three dimensional titanium miniplate in treatment of mandibular angle fracture"--a randomized prospective study. J Craniomaxillofac Surg. 2013 Mar;41(2):103-9. doi: 10.1016/j.jcms.2012.05.015. Epub 2012 Jul 17. PMID 22809633
- [Background] Farmand M, Dupoirieux L. [The value of 3-dimensional plates in maxillofacial surgery]. Rev Stomatol Chir Maxillofac. 1992;93(6):353-7. French. PMID 1475603
- [Background] Sadhwani BS, Anchlia S. Conventional 2.0 mm miniplates versus 3-D plates in mandibular fractures. Ann Maxillofac Surg. 2013 Jul;3(2):154-9. doi: 10.4103/2231-0746.119231. PMID 24205475
- [Background] Jain MK, Manjunath KS, Bhagwan BK, Shah DK. Comparison of 3-dimensional and standard miniplate fixation in the management of mandibular fractures. J Oral Maxillofac Surg. 2010 Jul;68(7):1568-72. doi: 10.1016/j.joms.2009.07.083. Epub 2010 Apr 22. PMID 20417012